CLINICAL TRIAL: NCT06840899
Title: Cannabinoid Modulation for Neurogenic Lower Urinary Tract Dysfunction in Spinal Cord Injury
Brief Title: CBD for Lower Urinary Tract Dysfunction in Spinal Cord Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0012; A539800 (Other: UW Madison); SMPH/UROLOGY/UROLOGY (Other: UW Madison); Protocol Version 9/16/24 (Other: UW Madison)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Supra-sacral Spinal Cord Injury; Spinal Cord Injury; Urinary Incontinence
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Incontinence | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBD for urinary incontinence (Experimental): Participants will take CBD for 90 days
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD — Twice daily 100mg cannabidiol (CBD)
  Other Names: Epidiolex

SUMMARY:
The goal of this feasibility study is to learn whether Cannabidiol (CBD) can improve urinary incontinence and other symptoms in people with recent spinal cord injury (SCI).

Participants will take Epidiolex (purified CBD) for 90 days

DETAILED DESCRIPTION:
This pilot study assesses the feasibility of using 100mg of twice daily cannabidiol (Epidiolex) in adult spinal cord injury with neurogenic lower urinary tract dysfunction following resolution of spinal shock.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* History of supra-sacral spinal cord injury of any mechanism
* Urinary incontinence with ≥2 episodes of urinary incontinence per day (outside of spinal shock)
* Willingness to participate in drug intervention trial
* English-speaking (able to provide consent and complete questionnaires)

Exclusion Criteria:

* History of intravesical Botox
* Actively taking >15 mg of Oxybutynin single dose or equivalent dose of alternative anticholinergic medication for bladder symptoms
* Use of Cannabis (any form) outside of study as determined by urine drug screen after washout period of 1 month if prior Cannabis use reported
* Thought or mood disorder aside from depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adherence to CBD (Epidiolex) regimen | 90 days
  Participants will complete a daily smartphone application-based drug diary recording when they take study drug.
Completion of 72-hour voiding diary | 90 days
  This assessment involves electronic participant documentation of urinary episodes at home.
Number of adverse events | 120 days
  Participants will be followed for adverse events for at least 30 days after the last dose of study drug.

SECONDARY OUTCOMES:
Change in urinary incontinence (UI) episodes | Baseline to 90 days
  Measured in the 72-hour voiding diary, participant documentation of urinary episodes at home.
Change in symptoms associated with UI | Baseline to 90 days
  Measured on 72-hour voiding diary, participant documentation of urinary episodes at home.
Change in urinary symptoms associated with neurogenic bladder | Baseline to 90 days
  Measured using Neurogenic Bladder Symptom Score - Short Form (NGBSS-SF). NGBSS-SF is a 10 question survey assessing the following domains: bladder management strategy, incontinence, storage & voiding, consequences, and quality of life. The total score ranges from 0 (no symptoms) to 28 (most severe symptoms). A higher total score indicates greater severity of neurogenic bladder symptoms.

OTHER OUTCOMES:
Change in Urodynamics - bladder capacity | Baseline to 3 months
  Bladder capacity assessment will be performed using pressure sensing urinary and rectal catheters during bladder filling with a solution of saline and iodinated contrast (and emptying if able) with fluoroscopic assessment. This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - maximum detrusor pressure | Baseline to 3 months
  Max detrusor pressure assessment (cm H20) during bladder storage will be performed using pressure sensing urinary and rectal catheters during bladder filling with a solution of saline and iodinated contrast with fluoroscopic assessment. This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - bladder compliance | Baseline to 3 months
  Bladder compliance assessment (mL/cm H20) will be performed using pressure sensing urinary and rectal catheters during bladder filling with a solution of saline and iodinated contrast (and emptying if able) with fluoroscopic assessment. This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - neurogenic detrusor overactivity (NDO) episodes | Baseline to 3 months
  NDO episode (involuntary, sudden contractions of the bladder muscle leading to a strong urge to urinate and potentially causing urine leakage) assessment will be performed using pressure sensing urinary and rectal catheters during bladder filling with a solution of saline and iodinated contrast with fluoroscopic assessment. This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - urine leaks | Baseline to 3 months
  Urine leak assessment will be performed using fluoroscopy during bladder filling with a solution of saline and iodinated contrast. This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - vesicoureteral reflux | Baseline to 3 months
  Vesicoureteral reflux assessment will be performed using fluoroscopy during bladder filling with a solution of saline and iodinated contrast. This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - bladder neck appearance | Baseline to 3 months
  Bladder neck appearance assessment will be performed using fluoroscopic assessment during bladder filling with a solution of saline and iodinated contrast (and emptying or leak if present). This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - bladder shape | Baseline to 3 months
  Bladder shape assessment will be performed using fluoroscopy during bladder filling with a solution of saline and iodinated contrast. This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Urodynamics - presence of detrusor sphincter dyssynergia | Baseline to 3 months
  Presence of detrusor sphincter dyssynergia assessment will be performed using pressure sensing urinary and rectal catheters, electromyography, and fluoroscopy during bladder filling with a solution of saline and iodinated contrast (and emptying or leaking if present). This assessment will only be completed for the first 10 participants to complete 3 months of treatment.
Change in Brief Pain Inventory (BPI) | Baseline to 3 months
  BPI is a 9 item survey assessing pain severity and impact on quality of life. Participants rate their pain on a scale of 0 to 10, where 10 is the worst pain imaginable. Participants also rate how much the pain interferes with their daily life on a scale of 0 to 10, where 10 is complete interference. Total combined range is 1-10, where pain severity and interference are: Mild: A score of 1-4; Moderate: A score of 5-6; and, Severe: A score of 7-10.
Change in Neurogenic Bowel Dysfunction Score (NBD) | Baseline to 3 months
  NBD is a 10 item system used to assess the severity of bowel dysfunction in individuals with neurological conditions, typically caused by spinal cord injuries, by assigning points based on the frequency and severity of symptoms like bowel movements, incontinence, and discomfort during defecation; a higher score indicates more severe neurogenic bowel dysfunction. The 10-items are scored on an ordinal scale. The NBD weighted score ranges between 0 and 47 points. A higher overall NBD score indicates more severe bowel symptoms. Score 0-6: Very minor; Score 7-9: Minor; Score 10-13: Moderate; and, Score 14+: Severe
Change in Pittsburgh Sleep Quality Index (PSQI) Questionnaire | Baseline to 3 months
  PSQI is a 19 item questionnaire assessing quality of sleep. Each component score ranges from 0 to 3, with 3 indicating the most disturbance. Total score is a number between 0 and 21 that indicates how well someone sleeps. A higher score means worse sleep quality.
Patient Global Impression Scale (PGI-C) | 3 months
  The PGI-C is a single question survey assessing change in overall clinical status after intervention. Answers range from Very much improved to Very much worse.
Change in International Spinal Cord Injury Quality of Life Basic Data Set (SCI QOL) | Baseline, 3 months, and 4 months
  The SCI QOL is a 3-item questionnaire to assess quality of life after spinal cord injury. It is scored on a 10 point Likert scale, with an overall range of 0-30. Lower scores indicate lower satisfaction with quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Javi Santiago, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes